CLINICAL TRIAL: NCT00812344
Title: An Open, Randomised, Cross-over, Single Centre Pharmacokinetic (Phase I) Study of the Biliary Excretion Following Single Doses of AZD0837, Given in the Duodenum Via a Loc-I-Gut Catheter, Alone or in Combination With Ketoconazole (Once Daily for 4 Days), to Young Healthy Male Subjects
Brief Title: Effect of Ketoconazole on Biliary Excretion of AZD0837
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Karin Wåhlander, MSD, AstraZeneca R&D Mölndal
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: D1250C00029
Record Dates: First submitted 2008-12-19; First posted 2008-12-22 (Estimated); Last update posted 2010-12-03 (Estimated); Status verified 2010-12

CONDITIONS: Healthy
Keywords: pharmacokinetics
MeSH Terms: interventions — AZD 0837; Ketoconazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: AZD0837
- 2 (Active Comparator): AZD0837 + Ketoconazole
  Interventions: Drug: AZD0837; Drug: Ketoconazole

INTERVENTIONS:
Drug: AZD0837 — Oral solution, dosing through the Loc-I-Gut catheter, single dose
Drug: Ketoconazole — tablets, orally, once daily for 3 days
  Arms: 2
Drug: ketoconazole — dissolved tablets, dosing through the Loc-I-Gut catheter, single dose
  Arms: 2

SUMMARY:
This is an explorative study and the scientific question to be investigated is if the biliary excretion of AZD0837 and its metabolites AR-H069927XX and AR-H067637XX are affected by co-administration with ketoconazole

ELIGIBILITY:
Inclusion Criteria:

* body mass index (BMI) between 19 to 30 kg/m2 and body weight between 50 to 100 kg inclusive

Exclusion Criteria:

* Significant illness, trauma or surgical procedures.
* Clinically significant laboratory abnormalities.
* Clinically significant medical history

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2008-12; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Amount of AZD0837, AR-H069927XX, and AR-H067637XX in bile and biliary clearance of AZD0837, AR-H069927XX, and AR-H067637XX. | Frequent sampling through a Loc-I-Gut catheter for up to 3 hours post dose.

SECONDARY OUTCOMES:
PK variables of AZD0837, AR-H069927XX, and AR-H067637XX. | Frequent sampling during 24 hours.
Adverse events, physical examination, safety laboratory variables, blood pressure, pulse and electrocardiography. | Some of the safety variables will be followed at each visit, some less frequent.
Pharmacogenetics | One sampling during the study.

CONTACTS AND LOCATIONS:
Overall Officials: Lars Knutson, MD, PhD, Principal Investigator — Inst för Kirurgiska VetenskaperUppsala Universitet
Locations (1):
- Research Site, Uppsala, Sweden